CLINICAL TRIAL: NCT04497428
Title: Brain Structures in Speech Motor Memory Consolidation
Brief Title: Sensory Basis of Speech Motor Learning
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: Yale University (Other)
Collaborators: McGill University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025475; R01DC017439 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Speech; Consolidation
MeSH Terms: conditions — Speech | interventions — Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adaptation to Altered Sensory Feedback + cTBS to S1 (Experimental): Adaptation to Altered Sensory Feedback + cTBS to S1
  Interventions: Behavioral: Adaptation; Other: cTBS
- Adaptation to Altered Sensory Feedback + cTBS to A1 (Experimental): Adaptation to Altered Sensory Feedback + cTBS to A1
  Interventions: Behavioral: Adaptation; Other: cTBS
- Adaptation to Altered Sensory Feedback + cTBS to M1 (Experimental): Adaptation to Altered Sensory Feedback + cTBS to M1
  Interventions: Behavioral: Adaptation; Other: cTBS
- Adaptation to Altered Sensory Feedback + Sham cTBS (Experimental): Adaptation to Altered Sensory Feedback + Sham cTBS
  Interventions: Behavioral: Adaptation; Other: cTBS

INTERVENTIONS:
Behavioral: Adaptation — Sensorimotor adaptation in speech
Other: cTBS — continuous theta-burst stimulation

SUMMARY:
These studies test the hypothesis that sensory areas of the brain participate in the consolidation of speech motor memory by using transcranial magnetic stimulation to suppress activity in somatosensory and auditory cortex following adaptation in order to block retention of learning.

DETAILED DESCRIPTION:
Subjects will train using either altered somatosensory feedback or altered auditory feedback (different groups of subjects). Immediately following adaptation, continuous theta burst magnetic stimulation (cTBS) will be applied to either auditory or somatosensory or motor cortex with the goal of blocking consolidation of motor memory. The logic of applying cTBS to both sensory areas is to test the hypothesis that both areas are involved in motor memory consolidation. Subjects leave the laboratory following cTBS and return 24 hours later to assess retention of learning. Learning is assessed as percentage change in speech sounds or movements relative to baseline. Retention is measured on a 0 to 100 scale relative to the end of learning.

ELIGIBILITY:
Inclusion Criteria:

* right handed adults
* no known physical or neurological abnormalities

Exclusion Criteria:

* patients with:
* cardiac pacemaker
* surgical clips or values on the heart
* implants
* metal or metallic fragments in any part of the body
* pregnancy
* claustrophobia
* a personal or family history of epilepsy
* currently taking antipsychotic drugs
* currently taking antidepressant drugs
* currently taking antianxiety drugs
* history of concussion.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Motor Learning | Performance as measured at the end of learning (30 minute session)
  Learning is assessed as percentage change in speech sounds (speech formant frequencies) or movements (movement curvature) relative to baseline.
Retention of Learning | 24 hours after learning (re-test lasts 30 minutes)
  Retention is measured on a 0 to 100 scale relative to the end of learning.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Haskins Laboratories
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT04497428/ICF_000.pdf